CLINICAL TRIAL: NCT02483052
Title: A Prospective Study of RejuvenAir System Radial Spray Cryotherapy to Determine Safety and Delayed Histological Effect in the Lung
Brief Title: RejuvenAir Lobectomy for Safety and Histology
Acronym: LobectomyCAN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CSA Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 013
Record Dates: First submitted 2015-06-24; First posted 2015-06-26 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Lung Neoplasms; Pulmonary Neoplasms
Keywords: lobectomy; spray cryotherapy; lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: RejuvenAir
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RejuvenAir (Experimental): RejuvenAir if the treatment areas are designated as Segmental, males will be dosed for 11 seconds and females for 10 seconds. If dosing is in the Lobar area males will be dosed for 12 seconds and females for 11 seconds.
  Interventions: Device: RejuvenAir

INTERVENTIONS:
Device: RejuvenAir — RejuvenAir
  Other Names: RejuvenAir™ System Radial Spray Cryotherapy

SUMMARY:
RejuvenAir System treatment will be performed during preoperative bronchoscopy 2 to 90 days prior to prescheduled lung resection in Subjects requiring lobectomy for removal of peripheral tumors. Treatment will be limited to areas of the bronchi within the lobe that will be removed, distal to the anticipated margin of resection. Treatment should be at least 1 cm from the bronchial resection margins and away from the tumor bed. Treated airways will be inspected via bronchoscopy at the time of thoracotomy, and examined histologically following surgical resection. Subject participation will be from 1 to 90 days and enrollment is anticipated to take 3 months. Subject having a RejuvenAir procedure and not going on to a resection for any reason will be followed for a maximum of 90 days for safety and undergo bronchoscopic evaluation of the treated airways at 90 days (+/- 4 Days)) post treatment.

DETAILED DESCRIPTION:
The study is a prospective, open label, single arm, single center study. The objective is to study the safety of the RejuvenAir System in a population of subjects who are scheduled to undergo a planned lobectomy. A secondary objective is to determine the histological effects of RejuvenAir System treatment in the airways. The Primary Endpoint is Safety as measured by occurrence of serious adverse events related to metered dose radial spray cryotherapy treatment performed prior to scheduled lobectomy surgery. The patient population intended to participate in this study are subjects scheduled to undergo lobectomy for peripheral lung lesions suspicious for or known to be cancer. Secondarily, this will enable an understanding of the histological characteristics and healing outcomes post-treatment in the airways, which will be resected. CSA Medical has conducted bench and animal studies that support the use of the RejuvenAir System as sufficiently safe and effective to warrant advancing the product into this primary safety study in patients presenting for consideration of lobectomy. Such patients provide a safe population to further the clinical evaluation of the system in that these subjects will receive their lobectomy or procedure 2 to 14 days following delivery of their metered liquid nitrogen treatment. At the time of their metered liquid nitrogen treatment they will be in an operating room setting with their thoracic surgeon in attendance. It is anticipated that subjects who agree to participate in this study will have the metered liquid nitrogen treatment at the time of evaluation of their lung lesion. This evaluation will include bronchoscopy with ultrasound for evaluation of their lymph nodes prior to the planned surgical resection of their lung abnormality.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of 21 to 75 years of age.

  * Subject is able to read, understand, and sign a written Informed Consent to participate in the study.
  * Subject is scheduled within 90 days from date of study treatment for a lobectomy unrelated to this study (upper and lower lobes only). Preferred range is 2-14 days from study treatment.
  * Subject has a pre-procedure post bronchodilator FEV1 of greater than or equal to 40% of predicted.
  * Subject is able to undergo bronchoscopy in the opinion of the investigator or per hospital guidelines.
  * Subject is able to adhere to and undergo a scheduled bronchoscope procedure prior to their clinically scheduled lobectomy surgical procedure.

Exclusion Criteria:

* • Subject is pregnant, nursing, or planning to get pregnant during study duration.

  * Subject is scheduled to have a pneumonectomy or has had a previous contralateral pneumonectomy.
  * Subject has had prior radiation therapy which involved the lungs.
  * Subject has received chemotherapy within the past 6 months, or is anticipated to be treated with chemotherapy between initial study treatment and lobectomy procedure.
  * Subject has an acute pulmonary infection or pneumonia within 6 weeks prior to study bronchoscopy.
  * Subject has had COPD exacerbation within 6 weeks prior to study bronchoscopy.
  * Subject has bronchiectasis in the area to be treated.
  * Subject has bullous emphysema. Characterized as large bullae >3 centimeters and confirmed on CT.
  * Subject has had a Lung transplant.
  * Subject has had lung reduction surgery, including implanted emphysema stent (s) implanted, coils or other devices for treatment.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Safety measured by occurrence of serious adverse events related to metered dose radial spray cryothreapy | prior to lobectomy-up to 14 days

SECONDARY OUTCOMES:
Histology assessed by description of depth of histological treatment effect per specified treatment dose | up to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Kashif Irshad, MDCM, MSc, Principal Investigator — WIlliam Osler Health Systems
Locations (1):
- William Osler Health System, Brampton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No